CLINICAL TRIAL: NCT02523599
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study to Investigate the Efficacy and Safety of the XaraColl® Bupivacaine Implant (300 mg Bupivacaine Hydrochloride) After Open Laparotomy Hernioplasty
Brief Title: Phase 3 Study of Efficacy and Safety of the XaraColl® Bupivacaine Implant After Hernioplasty
Acronym: MATRIX-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Innocoll (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INN-CB-014
Record Dates: First submitted 2015-08-12; First posted 2015-08-14 (Estimated); Results first posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Pain, Postoperative
Keywords: post operative pain; hernioplasty; bupivacaine
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- XaraColl (Experimental): 3 XaraColl Bupivacaine Implants each containing 100 mg of bupivacaine hydrochloride, for a 300 mg total dose
  Interventions: Drug: XaraColl
- Placebo (Placebo Comparator): 3 placebo implants
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: XaraColl — Surgical implantation of 3 bupivacaine collagen implants
  Other Names: Bupivacaine collagen implant
  Arms: XaraColl
Other: Placebo — Plain collagen implant (vehicle)
  Arms: Placebo

SUMMARY:
This is a Phase 3, multicenter, randomized, double-blind, parallel-group, placebo-controlled efficacy and safety study of postoperative pain in adults who are scheduled for unilateral inguinal hernioplasty via open laparotomy (tension-free technique).

Patients will assess their postoperative pain intensity (PI) using an 11-point numerical rating scale (NRS) from 0 hour through 72 hours postoperatively.

The expected maximum study duration for each patient will be up to 60 days, including a maximum 30-day screening period, the day of surgery and implantation, and a 30-day post implantation period including treatment and follow-up.

DETAILED DESCRIPTION:
This is a Phase 3, multicenter, randomized, double-blind, parallel-group, placebo-controlled study in adults who are scheduled for unilateral inguinal hernioplasty via open laparotomy (tension-free technique). Patients will receive either 3 XaraColl Bupivacaine Implants each containing 100 mg of bupivacaine hydrochloride, for a 300 mg total dose; or 3 placebo-sponges.

Three test article sponges will be implanted according to the patient's blinded treatment assignment. Following surgery, patients will be transferred to a postanesthesia care unit (PACU) and/or other postoperative recovery area for observation where they may receive parenteral morphine as needed (rescue medication for breakthrough pain) and on request for pain control. Once patients can tolerate oral medication, they will commence a standardized oral analgesic regimen with additional PRN medication to manage breakthrough pain only when it occurs.

Patients will assess their postoperative pain intensity (PI) using an 11-point numerical rating scale (NRS) from 0 hour through 72 hours postoperatively.

Patients will be observed postoperatively for a minimum of 3 hours and may be discharged at any time following completion of their 3-hour vital sign and PI assessments. Patients will be contacted at approximately 6, 24 and 48 hours after implantation to ensure protocol compliance and to perform safety assessments (including AEs and concomitant medications). At 72 hours, patients will return to the clinic to perform their final PI assessment, complete a categorical assessment of their overall pain control, and for follow-up safety assessments. They will also be asked to record the incidence of any ongoing or subsequent AEs (and any associated treatment) through Day 7. Additional follow-up assessments for safety will be performed at postoperative Day 7 (telephone call) and Days 15 and 30 (clinic visits).

ELIGIBILITY:
Inclusion Criteria:

* Has a planned (non-emergent) unilateral inguinal hernioplasty (open laparotomy, tension-free technique) to be performed according to standard surgical technique under general anesthesia. Repair of multiple hernias through a single incision is permitted provided only a single mesh will be used.
* If female, is nonpregnant and nonlactating.
* If female, is either not of childbearing potential (defined as postmenopausal for ≥ 1 year or surgically sterile [bilateral tubal ligation, bilateral oophorectomy or hysterectomy]) or practicing 1 of the protocol specified medically-acceptable methods of birth control and agrees to continue with the regimen throughout the duration of the study:
* Has the ability and willingness to comply with the study procedures and use of the eDiary.
* Is willing to use only permitted medications throughout the study.
* Is willing to use opioid analgesia.
* Must be able to fluently speak and understand either English or Spanish and be able to provide meaningful written informed consent for the study.

Exclusion Criteria:

* Has a known hypersensitivity to amide local anesthetics, morphine, acetaminophen or bovine products.
* Is scheduled for bilateral inguinal hernioplasty or other significant concurrent surgical procedures per investigator discretion.
* Has undergone major surgery within 3 months of the scheduled hernioplasty or plans to undergo another laparotomy procedure within 30 days postoperatively.
* Has used any analgesic other than acetaminophen within 24 hours of surgery. Acetaminophen may be used on the day of surgery but is subject to preoperative restrictions for oral intake.
* Has used aspirin or aspirin-containing products within 7 days of surgery. Aspirin at a dose of ≤ 325 mg is allowed for cardiovascular prophylaxis if the patient has been on a stable dose regimen for ≥ 30 days before Screening.
* Has used systemic steroids, anticonvulsants, antiepileptics, antidepressants for the management of chronic pain, or monoamine oxidase inhibitors on a regular basis within 10 days of surgery.
* Has used any opioid analgesic for an extended daily basis (30 - 60 mg oral morphine equivalent per day for 3 or more days a week) within 4 weeks before surgery. Patients who, in the investigator's opinion, may be developing opioid tolerance are also excluded.
* Has any chronic painful condition (eg, fibromyalgia) or routinely uses pain medication other than acetaminophen (including nonsteroidal anti-inflammatory drugs [NSAIDs]) that, in the opinion of the investigator, may confound the assessment of pain associated with the hernioplasty.
* Has a physical or mental condition that, in the opinion of the investigator, may confound the assessment of postoperative pain after hernioplasty.
* Shows evidence of tolerance or physical dependency on opioid analgesics or sedative-hypnotic medications.
* Has a urine drug screen that tests positive for drugs of abuse or misuse, including cannabinoids.
* Has liver function test results greater than 3x the upper limit of normal or a history of cirrhosis.
* Has any clinically significant unstable cardiac disease (eg, uncontrolled hypertension, clinically significant arrhythmia at baseline, or an implantable cardioverter-defibrillator [ICD])
* Has any clinically significant unstable neurological, immunological, renal, or hematological disease (eg, uncontrolled diabetes or significantly abnormal laboratory findings), or any other condition that, in the opinion of the investigator, could compromise the patient's welfare, ability to communicate with the study staff or otherwise contraindicate study participation.
* Has an open workman's compensation claim.
* Has participated in a clinical trial (investigational or marketed product) within 30 days of surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2015-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn Niebler, D.O., Study Director — Innocoll
Locations (21):
- United States (21):
  - Mobile, Alabama
  - Sheffield, Alabama
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Encino, California
  - Bradenton, Florida
  - Clermont, Florida
  - Inverness, Florida
  - Kissimmee, Florida
  - Miami, Florida
  - Orlando, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Weston, Florida
  - Indianapolis, Indiana
  - Springfield, Massachusetts
  - Flint, Michigan
  - Las Vegas, Nevada
  - El Paso, Texas
  - Houston, Texas
  - Lampasas, Texas

REFERENCES:
- [Derived] Velanovich V, Rider P, Deck K, Minkowitz HS, Leiman D, Jones N, Niebler G. Safety and Efficacy of Bupivacaine HCl Collagen-Matrix Implant (INL-001) in Open Inguinal Hernia Repair: Results from Two Randomized Controlled Trials. Adv Ther. 2019 Jan;36(1):200-216. doi: 10.1007/s12325-018-0836-4. Epub 2018 Nov 22. PMID 30467808

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | XaraColl | Placebo
Started | 204 | 101
Randomized But Not Treated | 1 | 0
Completed | 196 | 100
Not Completed | 8 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 4 | 1
Not completed — Did not return for Day 30 visit | 2 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat
Groups:
- Total: Total of all reporting groups
Arm/Group | XaraColl | Placebo | Total
Number analyzed (Participants) | 204 | 101 | 305
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (12.82) | 53.3 (14.01) | 53.1 (13.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 196 | 97 | 293
Region of Enrollment [Number; unit: participants]
  United States | 204 | 101 | 305

OUTCOME MEASURES:

1. Primary Outcome: SPI24
Description: Sum of Pain Intensity (SPI24). The time weighted sum of pain intensity from 0 to 24 hours (ie, the area under the NRS PI curve from 0 to 24 hours). Where 0 indicated "no pain" and 10 indicated "worst pain possible". This type of measurement scale is called "NRS" or Numerical Rating Scale For the purpose of (SPI) computation, PI at Time 0 (Baseline PI) is set to zero for all patients who have test article implantation. SPI will not be calculated for randomized but not treated patients. A lower score is a better outcome. Minimum value would be "0" and Maximum value would be 240. Time-weighted SPI is calculated as the sum of the pain intensities between successive time points (i.e., if SPI24 = ∑[PI x (time t - time t-1)], where "t" represents a given time point,"t-1" represents the previous time point, and time is expressed in hours). This represents the AUC (Area Under the Curve) of the pain intensities when calculated with the trapezoidal rule.
Time Frame: 0 to 24 hours
Population: mITT Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | XaraColl | Placebo
Number analyzed (Participants) | 197 | 101
units on a scale | 85.0 (47.18) | 106.8 (48.20)

2. Secondary Outcome: TOpA24
Description: Total use of opioid analgesia (TOpA) from Time 0 through 24 hours (TOpA24). This is a basic measurement of counting in total the number of morphine tablets (15 mg) patients had use within a 24 hour period (typically called "rescue" to help manage pain. Zero (0) is the "lowest" score. The lower the number of tablets the better outcome.
Time Frame: Time 0 through 24 hours
Population: (mITT Population)
Measure: Median (95% Confidence Interval); unit: morphine mg equivalent
Arm/Group | XaraColl | Placebo
Number analyzed (Participants) | 197 | 101
morphine mg equivalent | 5 [0 to 47] | 10 [0 to 40]

3. Secondary Outcome: TOpA48
Description: Total use of Opioid Analgesia from Time 0 through 48 hours (TOpA48) This is a basic measurement of counting in total the number of morphine tablets (15 mg) patients had use within a 48-hour period (typically called "rescue" to help manage pain. Zero (0) is the "lowest" score. The lower the number of tablets the better outcome.
Time Frame: Time 0 through 48 hours
Population: mITT Population
Measure: Median (95% Confidence Interval); unit: morphine mg equivalent
Arm/Group | XaraColl | Placebo
Number analyzed (Participants) | 197 | 101
morphine mg equivalent | 5.0 [0.0 to 82.0] | 14.0 [0.0 to 65.0]

4. Secondary Outcome: TOpA72
Description: Total use of Opioid Analgesia (TOpA) from Time 0 through 72 hours. This is a basic measurement of counting in total the number of morphine tablets patients had use within a 72-hour period (typically called "rescue" to help manage pain. Zero (0) is the "lowest" score. The lower the number of tablets the better outcome.
Time Frame: Time 0 through 72 hours
Measure: Median (95% Confidence Interval); unit: morphine mg equivalent
Arm/Group | XaraColl | Placebo
Number analyzed (Participants) | 197 | 101
morphine mg equivalent | 5.0 [0.0 to 102.0] | 14.0 [0.0 to 100.0]

5. Secondary Outcome: SPI48
Description: Sum of pain intensity (SPI).The time weighted sum of pain intensity from 0 to 48 hours (ie, the area under the NRS PI curve from 0 to 48 hours). For the purpose of SPI computation, Pain Intensity at Time 0 (Baseline PI) is set to zero for all patients who have test article implantation. Minimum value would be "0" and Maximum value would be 480. Time-weighted SPI is calculated as the sum of the pain intensities between successive time points (i.e., if SPI24 = ∑[PI x (time t - time t-1)], where "t" represents a given time point,"t-1" represents the previous time point, and time is expressed in hours). This represents the AUC (Area Under the Curve) of the pain intensities when calculated with the trapezoidal rule.
Time Frame: 0 to 48 hours
Population: mITT Population
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | XaraColl | Placebo
Number analyzed (Participants) | 197 | 101
units on a scale | 165.7 [0.0 to 408.9] | 190.1 [6.6 to 470.7]

6. Secondary Outcome: SPI72
Description: Sum of pain intensity (SPI). The time weighted sum of pain intensity from 0 to 72 hours (ie, the area under the NRS PI curve from 0 to 72 hours). For the purpose of SPI computation, PI at Time 0 (Baseline PI) is set to zero for all patients who have test article implantation. Where 0 indicates "no pain" and 10 indicated "worst pain possible". A lower score is a better outcome. Minimum value would be "0" and Maximum value would be 720. Time-weighted SPI is calculated as the sum of the pain intensities between successive time points (i.e., if SPI72 = ∑[PI x (time t - time t-1)], where "t" represents a given time point,"t-1" represents the previous time point, and time is expressed in hours). This represents the AUC (Area Under the Curve) of the pain intensities when calculated with the trapezoidal rule.
Time Frame: 0 to 72 hours
Population: mITT Population
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | XaraColl | Placebo
Number analyzed (Participants) | 197 | 101
units on a scale | 245.2 [0.0 to 594.1] | 263.3 [6.6 to 710.4]

ADVERSE EVENTS:
Time Frame: 30 days
Description: A total of 204 patients have been randomized to INL-001 active drug arm. However 1 patient was randomized and not treated. This means only 203 patients received the active compound. In the Placebo arm all patient randomized were treated.
Arm/Group | XaraColl | Placebo
Serious Adverse Events (participants affected / at risk) | 2/203 | 0/101
Other Adverse Events (participants affected / at risk) | 103/203 | 55/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XaraColl (N=203) | Placebo (N=101)
intestinal ischemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
sepsis (Infections and infestations) | 1 (1) | 0 (0)
peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XaraColl (N=203) | Placebo (N=101)
constipation (Gastrointestinal disorders) | 17 (17) | 12 (12)
nausea (Gastrointestinal disorders) | 23 (23) | 15 (15)
incision site pain (Injury, poisoning and procedural complications) | 34 (34) | 19 (19)
incision site swelling (Injury, poisoning and procedural complications) | 42 (42) | 19 (19)
post procedural discharge (Injury, poisoning and procedural complications) | 15 (15) | 6 (6)
dizziness (Nervous system disorders) | 31 (31) | 12 (12)
dysgeusia (Nervous system disorders) | 14 (14) | 3 (3)
somnolence (Nervous system disorders) | 36 (36) | 20 (20)
restlessness (Psychiatric disorders) | 14 (14) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other